CLINICAL TRIAL: NCT02331290
Title: Excretion of Acetylamantadine (AA) by Lung Cancer Patients During a Chemotherapy Regimen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: CancerCare Manitoba (Other)
Responsible Party: Sponsor
Other Study IDs: RRIC 2014-047
Record Dates: First submitted 2014-11-05; First posted 2015-01-06 (Estimated); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood (2 x 10 ml) at 2 and 4 hours after amantadine ingestion. Saliva (2 x 5ml) immediately after the blood samples. Urine specimen between the time of the 2 blood samples.
  The sampling protocol will be repeated 3 weeks later with the second cycle of chemotherapy.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: 20 newly diagnosed patients with small-cell lung cancer and adenocarcinoma of the lung stage III or IV

SUMMARY:
This study is designed to determine if changes in acetyl amantadine (AA) metabolism with systemic chemotherapy - reflective of SSAT1 activity - are predictive of response to systemic therapy in patients with lung cancer. Ten patients with adenocarcinoma and 10 with small-cell cancer who are at American Joint Committee on Cancer (AJCC) stages 3 or 4 at the time of diagnosis will participate. AA metabolites will be examined by ELISA prior to initiation of systemic chemotherapy and after the second cycle of therapy. Changes in the pattern of metabolites will be correlated with convention clinical and radiographic response criteria.

DETAILED DESCRIPTION:
Evaluation of response to systemic therapy is dependant on clinical and radiographic changes assessed prior to and after several cycles of systemic therapy. The response rate for lung cancer to systemic therapy ranges from 30 - 85%, depending on histology and other clinical factors, but difficult to predict in individual patients. Spermine-spermidine acetyl transferase (SSAT1) activity is up-regulated in many cancers and may be a marker of response to therapy. Metabolism of acetyl amantadine (AA) is reflective of SSAT1 activity. In order to determine if change in SSAT1 activity is predictive of response to systemic chemotherapy, we propose the following pilot clinical trial. A total of 20 volunteer patients - 10 patients with adenocarcinoma of the lung and 10 patients with small-cell histology will be included. Eligibility includes patients with adenocarcinoma and small-cell lung cancer who are at AJCC stage III or IV at diagnosis. Volunteers will be informed that this study is examining the possibility that we can detect a therapeutic response by a change in their excretion of AA before it can be detected by conventional patient assessment methods. The chemotherapy regimen will be selected by the treating physician and will not be influenced by participation in this clinical trial. The usual treatment regimen for the entities described above is a platinum-based doublet, often cis-platin with etoposide or gemcitabine administered for 4 to 6 cycles. The therapeutic response rates with these drug regimens is about 40% for adenocarcinoma and 70% for small-cell carcinoma. Clinical response is usually assessed between the second and third cycles of chemotherapy.

Biological Sampling Details

Patient volunteers will be asked to fast overnight prior to the day of their first scheduled chemotherapy and to ingest an oral dose of 200 mg of amantadine hydrochloride (HCl) in the morning within an hour of arriving in clinic. The following biological specimens will be collected: blood (2 x 10 ml) at 2 and 4 hours after amantadine ingestion, saliva (2 x 5ml) immediately after the blood samples, and a total urine specimen between the time of the 2 blood samples. Patient will be instructed to empty the bladder immediately before the first blood sample and then collect the total urine produced until the end of the second blood sample (4 hours). Subsequently, the patient will be allowed lunch (if they so choose) prior to their scheduled chemotherapy.

The sampling protocol will be repeated 3 weeks later with the second cycle of chemotherapy.

Data to be collected: tumour type (histology), stage of cancer, age, sex, weight, height, smoking history, concurrent medications, systemic chemotherapy treatment prescribed and history of recent alcohol intake. Data will be used for correlation and to determine the relationship of plasma, salivary or urinary AA to the particular cancer diagnosis and response to treatment.

Primary Endpoints:

Documentation of acetylamantadine metabolite excretion/secretion.

Response to therapy (complete response, partial response, stable disease, progressive disease).

Time to disease recurrence or progression.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven newly diagnosed advanced-stage small-cell lung cancer (SCLC) and adenocarcinoma of the lung being initiated on systemic chemotherapy.
* Adequate hematological, renal and hepatic function sufficient to tolerate conventional doses of systemic chemotherapy.
* Age > 18 years.
* Measurable or evaluable disease by Response Evaluation Criteria in solid Tumors (RECIST) criteria.
* Performance score < 3 (ECOG).
* Capable of signing informed consent.

Exclusion Criteria:

* Patients with significant liver and kidney disease, chronic drug therapy other then oral contraceptives. Pregnant or lactating female patients.
* Women with childbearing potential must have a negative pregnancy test and be willing to use effective contraceptive techniques if sexually active.
* Previous history of adverse reactions to amantadine.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 patients: 10 patients with biopsy proven newly diagnosed Stage III or IV adenocarcinoma of the lung and 10 patients with Stage III or IV small-cell histology will be included.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Pattern of AA metabolite excretion/secretion relative to response to therapy. | Two months
  Correlation of AA metabolite excretion/secretion to response to systemic chemotherapy.

SECONDARY OUTCOMES:
Pattern of AA metabolite excretion/secretion relative to time to recurrence or progression. | Two years
  Correlation of AA metabolite excretion/secretion to time to disease recurrence or progression.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Maksymiuk, MD FRCP(C), Principal Investigator — CancerCare Manitoba
Locations (2):
- Canada (2):
  - St. Boniface Hospital, Winnipeg, Manitoba
  - CancerCare Manitoba, Winnipeg, Manitoba

REFERENCES:
- [Background] Bras AP, Janne J, Porter CW, Sitar DS. Spermidine/spermine n(1)-acetyltransferase catalyzes amantadine acetylation. Drug Metab Dispos. 2001 May;29(5):676-80. PMID 11302933